CLINICAL TRIAL: NCT04187547
Title: A Phase III, 26-Week, Double-blind, Randomised, Placebo-controlled, Parallel-group Trial to Investigate the Efficacy and Safety of Daily Administration of Tricaprilin as AC-SD-03 in Subjects With Mild to Moderately Severe Probable Alzheimer's Disease and Who Are Noncarriers of the APOE4 Allele
Brief Title: A Phase III Multi Regional Clinical Trial (MRCT) of Tricaprilin in Mild to Moderately Severe Probable Alzheimer's Disease With Optional Open Label Extension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study replaced with a new study
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-19-020
Record Dates: First submitted 2019-11-29; First posted 2019-12-05 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tricaprylin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AC-SD-03 (Active Comparator): Tricaprilin SD formulation, twice daily. Administered orally
  Interventions: Drug: Tricaprilin
- AC-SD-03P (Placebo Comparator): Placebo formulation, twice daily. Administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tricaprilin — Powder formulation will be mixed with 240 mL water and shaken until fully dispersed.
  Each dosing unit of AC-SD-03 contains 20 g of the active ingredients (tricaprilin)
  Other Names: AC-SD-03
  Arms: AC-SD-03
Drug: Placebo — Matching placebo to AC-SD-03 will be mixed with 240 mL water and shaken until fully dispersed.
  Other Names: AC-SD-03P
  Arms: AC-SD-03P

SUMMARY:
This is Phase 3 study, multi-centre, double-blind, placebo controlled, parallel group to evaluate the effects of AC-SD-03 on the efficacy and safety among participants with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 50 and 85 (inclusive) at the time of Screening Visit 1. Subjects 86 to 90 years of age (inclusive) can be enrolled, provided that the Medical Monitor reviews the subject's medical condition during the screening process and approves enrolment.
2. Dementia of mild to moderate severity, as classified by MMSE score between 14 to 26, inclusive, at Screening Visit 1.
3. Meets diagnostic clinical criteria of probable Alzheimer's dementia according to the National Institute on Aging and the Alzheimer's Association (NIA-AA) [25].
4. Magnetic resonance imaging prior to Visit 3 (Baseline) compatible with a diagnosis of probable AD.
5. Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) brain scan showing a pattern typical for AD according to central PET reader (with areas of glucose hypometabolism in posterior cingulate, temporal, parietal, and/or prefrontal cortices, as per criteria in imaging manual).
6. Confirmed APOE negative genotype result obtained by the central laboratory prior to Screening Visit 2 or documented prior to screening.
7. Subjects taking the following cholinesterase inhibitors (ChEI): donepezil, galantamine, or rivastigmine; and/or GV-971, and/or memantine and/or other agents which may impact cognition (e.g., Souvenaid®, NeuroAidTM, Cerefolin®, Gingko biloba, etc) are eligible for enrolment:

   1. If the subject has been taking such medication(s)/products for 3 months or more at Screening Visit 1.
   2. If the current dosage regimen is within the approved dose range.
   3. The daily dose has remained unchanged for at least 6 weeks prior to screening.
   4. If the dose is not expected to change during trial participation.
   5. Tacrine use is not allowed.
8. In the opinion of the Investigator, the subject's medical condition, except for dementia, has been stable for at least 3 consecutive months prior to Screening Visit 1.
9. Subjects do not have active suicidal thoughts (answers 'yes' to questions 4 or 5, on the Columbia-Suicide Severity Rating Scale [C-SSRS]) within 6 months preceding Screening Visit 2 or Visit 3 (Baseline). Additionally, subjects have no active history of suicide attempt in the previous 2 years or more than 1 lifetime suicide attempt, nor are they at serious suicidal risk, in the opinion of the Investigator.
10. The subject is able to comply with protocol testing and procedures for the entire length of the trial.
11. Has a permanent caregiver (subject's caregiver is not expected to change during the trial) who is willing to attend all visits, oversee the subject's compliance with protocol-specified procedures and IP administration, and report on subject's status. Caregiver must have, in the opinion of the Investigator, enough contact with the subject to be able to perform the duties described above.
12. The subject and caregiver are, in the Investigator's judgement, proficient in the language in which the trial assessments will be completed, and have hearing, vision and physical abilities adequate to perform assessments (corrective aids allowed).
13. Subject and caregiver must provide full written informed consent prior to the performance of any protocol-specified procedure; or if subject is unable to provide informed consent due to cognitive status, provision of informed consent by cognitively intact legally acceptable representative (where this is in accordance with local laws, regulations and ethics committee policy).
14. Subject is able to ingest oral medication.
15. Subject is able to tolerate a 5 g dose of tricaprilin (formulated as 12.5 g of AC-SD-03) as per sentinel dose challenge at Visit 3 (Baseline).

Exclusion Criteria:

1. Current use or use within 3 months of Visit 3 (Baseline), of Axona® or other MCT-containing products. Use of coconut oil up to 15 mL (1 tablespoon) per day is allowed. Use of MCT-containing products is not allowed at any time during trial participation.
2. Use of any other investigational agent within 60 days prior to Screening Visit 1.
3. Has a known allergy or hypersensitivity to triglycerides.
4. In the opinion of the Investigator, has presence or history of an advanced, severe, progressive, or unstable disease of any type that could interfere with efficacy and safety assessments, or put the subject at risk.
5. Has any medical or neurological condition, other than AD, that could explain the subject's dementia (e.g., structural abnormality, traumatic brain injury, stroke, epilepsy, Parkinson's disease, alcohol-related dementia, etc.)
6. Has a modified Hachinski Ischemia score greater than (>) 4 at Screening Visit 2.
7. Has a history or clinical laboratory evidence of cerebrovascular disease (stroke, transient ischemic attack, haemorrhage), or diagnosis of possible, probable, or definite vascular dementia at Screening Visit 1 in accordance with National Institute of Neurological Disorders and Stroke criteria.
8. Brain MRI performed at Screening (prior to Visit 3) (per centrally read MRI) that shows evidence of any of the following:

   1. Acute, sub-acute or chronic haemorrhage.
   2. Cortical infarct (defined as > 1.5 cm in diameter).
   3. > 1 lacunar infarct (defined as < 1.5 cm in diameter).
   4. Superficial siderosis.
   5. History of diffuse white matter disease as defined by a score of 3 on the age-related white matter changes scale [26].
   6. Any finding that, in the opinion of the Investigator, might be a contributing cause of subject's dementia, might pose a risk to the subject, or might prevent a satisfactory MRI assessment for safety monitoring.
9. Has a history or clinical laboratory evidence of moderate congestive heart failure defined by the New York Heart Association Criteria (Class I to IV).
10. Clinically significant ECG abnormalities at Screening Visit 2, for example:

    1. Evidence of atrial fibrillation on ECG or history of atrial fibrillation that is not currently controlled
    2. QTcF at > 450 ms in males or > 470 ms in females, or low or flat T waves making measurement of QT interval unreliable
11. Has a history of new ischemic or congestive cardiovascular event within the 3 months prior to Visit 3 (Baseline).
12. Has a history of or current major psychiatric illness such as schizophrenia or bipolar affective disorder.
13. Has a clinician-administered Patient Health Questionnaire (PHQ)-9 score of ≥ 10 or in the Investigator's opinion, depression of a severity that would impact cognitive assessments.
14. Subjects with insulin dependent diabetes.
15. Subjects with uncontrolled hypertension defined as:

    1. average of 3 systolic blood pressure [SBP]/diastolic blood pressure [DBP] readings > 165/100 mmHg at Screening Visit 2 (blood pressure measurements exceeding these limits may be repeated as warranted by the Investigator, but values must be within the specified limits for the subject to be eligible for the study),
    2. or persistent SBP/DBP readings > 180/100 mmHg 3 months prior to Baseline (Visit 3, Day 1) that in the opinion of the Investigator are indicative of chronic uncontrolled hypertension.
16. Subjects with orthostatic hypotension, defined as a drop of >20 mmHg systolic blood pressure upon standing upright from a seated position within 3 minutes, at Screening Visit 2; testing for orthostatic hypotension may be repeated at Investigator's discretion if there is reason to believe the condition is temporary after addressing the temporary cause.
17. At Screening Visit 2, clinically significant:

    1. anaemia (haemoglobin < 11 g/dL for males or < 10 g/dL for females)
    2. renal disease or insufficiency, including but not limited to a creatinine value of > 1.9 mg/dL (> 170 μmol/L)
    3. hypothyroidism
18. At Screening Visit 2, laboratory test values (potential to repeat at Investigators discretion):

    1. ALT, AST, total bilirubin, or alkaline phosphatase > 2.5 times the ULN laboratory range, or history of severe hepatobiliary disease (e.g., hepatitis B or C, or cirrhosis [Childs-Pugh Classes B/C] without enzyme elevation)
    2. Fasting triglycerides > 2.5 times the ULN
    3. Cholesterol > 240 mg/dL
19. Clinically significant Vitamin B12 deficiency within 12 months prior to Visit 1; however, subjects on stable replacement therapy for a minimum of 1 month immediately prior to Visit 1 may be included.
20. The following GI conditions are exclusionary as described below:

    1. Inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease), GI bleed (upper or lower), or peptic ulcer disease; any of these conditions are exclusionary, if active in the past 5 years. Subjects with remote quiescent disease, at Investigators discretion (and CER Committee) are not excluded.
    2. Subjects with current or a history of (within the last 5 years) any of the following conditions are excluded: complicated reflux disease (e.g., Barrett's oesophagus, stricture, ulcer, haemorrhage), or severe GERD that, in the opinion of the Investigator, is not well-controlled by medication.
    3. Irritable bowel syndrome, diverticular disease (e.g., diverticulosis, or diverticulitis), or chronic gastritis; any of these conditions are exclusionary if there has been an acute event within 1 year prior to Screening Visit 1.
21. Has donated ≥ 2 units of blood within the 1 month prior to Screening Visit 1.
22. Has a history of alcohol or drug abuse within the 6 months prior to Visit 1 or has tested positive upon urine drug screen at Screening Visit 2.
23. Subject or caregiver is an immediate family member or employee of the clinical site, Sponsor, or of the Sponsor's agents.
24. Has any current or history of neoplasm or malignancy, other than excised or treated basal cell carcinoma. The following exceptions may be made after discussion with the Medical Monitor:

    1. Subjects with cancers in remission more than 5 years prior to Screening.
    2. Subjects with a history of excised or treated squamous carcinoma of the skin.
    3. Subjects with prostate cancer in situ.
25. Subject has a scheduled (or is expected to have scheduled) hospitalisation and/or surgery during the trial

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Alzheimer's Disease Assessment Scale-cognitive Subscale (ADAS-cog11). Total Score up to 20-week Treatment | 20 weeks
  Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog 11) is an 11- item cognitive subscale that objectively measures memory, language, orientation, and praxis with a total score range of 0 (no impairment) to 70 (severe impairment).

SECONDARY OUTCOMES:
Number of subjects with treatment related adverse events | 20 weeks
  TEAE incidence rate per treatment group
Clinical Global Impression of Change | 20 weeks
  Clinician's global impression rated with Alzheimer's Disease cooperative Study - Clinical Global Impression of Change (ADCS-CGIC)
Change From Baseline in Dependence Scale.Total Score up to 20-week Treatment | 20 weeks
  The Dependence Scale is a 13-item scale with a total score from 0 to 15, where higher scores indicate more dependence.
Change From Baseline in RUD-Lite | 20 weeks
  The RUD-lite is an interview designed to assess resource utilisation required for subjects with dementia and their caregivers. Information gathered on both caregivers (caregiving time, work status) and participants (accommodation and healthcare resource utilization).
Change From Baseline in Disability Assessment for Dementia | 20 weeks
  The Disability Assessment for Dementia (DAD) is an interview designed to measure of functional ability in dementia.